CLINICAL TRIAL: NCT05713097
Title: Thyroid-stimulating Immunoglobulins Level in Patients With Graves' Disease Undergoing Maintenance-dose of Antithyroid Drug and Its Relationship With Disease Relapse
Brief Title: TSI and Its Relationship With Graves' Disease Relapse
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Phong VN Nguyen, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: TSI_Medic
Record Dates: First submitted 2023-01-13; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Graves Disease; Immunoglobulin; Anti-Thyroid Antibodies Disorder
Keywords: TSI; recurrent Graves' disease; Graves' ophthalmopathy; treatment duration; anti-thyroid drug; cut-off
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — TSI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATD withdrawal: ATD treatment was decided to be stopped at the discretion of the attending physician. Then, patients were followed after ATD withdrawal to determine who would have relapse of GD.
  Finally, patients were divided into 2 groups: Relapse and No relapse
  Interventions: Diagnostic Test: TSI
- No ATD withdrawal: Patients treated with ATD still the end of the study
  Interventions: Diagnostic Test: TSI

INTERVENTIONS:
Diagnostic Test: TSI — TSI was measured several times during the course of treatment when planning to stop medication (at the discretion of the attending physician).

SUMMARY:
The goal of this observational study is to determine the role of TSI, as well as clinical signs and thyroid function tests in predicting Graves' disease (GD) relapse after withdrawing anti thyroid drug (ATD). The main questions it aims to answer are:

1. To investigate the serum TSI concentration in patients with GD undergoing maintenance-dose ATD.
2. To determine an optimal cut-off of TSI level for predicting GD relapse.
3. To determine the role of TSI in predicting Graves' disease relapse after withdrawing ATD.

DETAILED DESCRIPTION:
Retrospective follow-up study of patients with hyperthyroidism due to Graves' disease, treated at the endocrine outpatient clinic of Medic Medical Center, Ho Chi Minh City from January 2000 to April 2021. TSI was measured several times during the course of treatment when planning to stop medication (at the discretion of the attending physician). ATD withdrawal would be planned when patients achieved euthyroid status clinically with normal FT4 tests for at least 3 months with minimal dose of ATD. The decision was also based on TSI concentration, goiter's characteristics and parenchymal vascularity on Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hyperthyroidism due to Graves' disease according to the criteria of the Japan Thyroid Association.
* TSI: measured during the course of treatment when planning to stop medication (normal FT4 at maintenance-dose of ATD) Methimazole (MMI): at doses of ≤10 mg. Propylthiouracil (PTU): at doses of ≤200 mg.

Exclusion Criteria:

* Hyperthyroidism due to other causes
* Patients who were intolerant to ATD or had serious side effects with ATD.
* TSIs were measured in pregnancy.
* Patients treated with surgery or radioactive iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hyperthyroidism due to Graves' disease, treated at the endocrine outpatient clinic of Medic Medical Center, Ho Chi Minh City, Vietnam from January 2000 to April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with GD relapse | at least 1 year after ATD withdrawal
  Patients who had relapse of hyperthyroidism due to GD

SECONDARY OUTCOMES:
TSI LEVEL IN PATIENTS WITH GRAVES' DISEASE UNDERGOING MAINTENANCE-DOSE OF ANTITHYROID DRUG. | before ATD withdrawal
  TSI level before planning for ATD withdrawal
Optimal cut-off of TSI level for predicting GD relapse | before ATD withdrawal
  Optimal cut-off of TSI level before ATD withdrawal for predicting GD relapse

CONTACTS AND LOCATIONS:
Overall Officials: Vu Nhat Phong Nguyen, MD, Principal Investigator — University of Medecine and Pharmacy at Ho Chi Minh City
Locations (1):
- Hoa Hao Clinic, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No